CLINICAL TRIAL: NCT02706262
Title: Complex Effects of Dietary Manipulation on Metabolic Function, Inflammation and Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PSQ-201512086
Record Dates: First submitted 2016-02-24; First posted 2016-03-11 (Estimated); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Insulin Resistance
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Metabolically normal lean - Baseline testing only (No Intervention): Metabolically normal lean - Lean individuals that have good glucose (sugar) control, normal plasma triglyceride (fat) levels and a low liver fat content.
  Dietary intervention - None.
- Metabolically normal obese - Baseline testing only (No Intervention): Metabolically normal obese - Persons with obesity that have good glucose (sugar) control, normal plasma triglyceride (fat) levels and a low liver fat content.
  Dietary intervention - None.
- Metabolically abnormal obese - Mediterranean diet (Experimental): Metabolically abnormal obese - Persons with obesity with glucose levels higher than recommended and a moderate to high amount of fat in the liver.
  Dietary intervention - A nutritionally balanced diet that includes fruits, vegetables, fish, beans, whole grains, and olive oil with approximately 50% of daily calories coming from complex carbohydrates, 30% of calories from fat, and 20% of calories from protein.
  Interventions: Other: Metabolically abnormal obese - Mediterranean diet; Behavioral: Annual Follow-up Visits
- Metabolically abnormal obese - Low carbohydrate ketogenic diet (Experimental): Metabolically abnormal obese - Persons with obesity with glucose levels higher than recommended and a moderate to high amount of fat in the liver.
  Dietary intervention - A very-low-carbohydrate, adequate protein, high-fat diet containing 20 grams of carbohydrate or less per day (about 5% of calories), derived mainly from vegetables.
  Interventions: Other: Metabolically abnormal obese - Low carbohydrate ketogenic diet; Behavioral: Annual Follow-up Visits
- Metabolically abnormal obese - Plant-based very-low-fat diet (Experimental): Metabolically abnormal obese - Persons with obesity with glucose levels higher than recommended and a moderate to high amount of fat in the liver.
  Dietary intervention - A plant-based diet high in complex carbohydrates and low in fat, protein, and sodium, with approximately 70% of daily calories from carbohydrates, 15% from fat, and 15% from protein.
  Interventions: Other: Metabolically abnormal obese - Plant-based, very-low-fat diet; Behavioral: Annual Follow-up Visits

INTERVENTIONS:
Other: Metabolically abnormal obese - Mediterranean diet — The effect of consuming a Mediterranean diet will be examined over 3 different phases: (i) weight maintenance for 4 to 8 weeks, with all meals provided; (ii) controlled 7-10% weight loss with caloric intake reduced by 25% to achieve the desired amount of weight loss in about 4 to 5 months with all meals provided; and (iii) Independent weight loss for about 4 months. During the independent weight loss phase of the study subjects will be asked to continue to consume a Mediterranean diet but will prepare all their food at home. No food will be provided during this portion of the study.
  Arms: Metabolically abnormal obese - Mediterranean diet
Other: Metabolically abnormal obese - Low carbohydrate ketogenic diet — The effect of consuming a low-carbohydrate, ketogenic diet will be examined over 3 different phases: (i) weight maintenance for 4 to 8 weeks, with all meals provided; (ii) controlled 7-10% weight loss with caloric intake reduced by 25% to achieve the desired amount of weight loss in about 4 to 5 months with all meals provided; and (iii) Independent weight loss for about 4 months. During the independent weight loss phase of the study subjects will be asked to continue to consume a low carbohydrate ketogenic diet but will prepare all their food at home. No food will be provided during this portion of the study.
  Arms: Metabolically abnormal obese - Low carbohydrate ketogenic diet
Other: Metabolically abnormal obese - Plant-based, very-low-fat diet — The effect of consuming a plant-based, very-low-fat diet will be examined over 3 different phases: (i) weight maintenance for 4 to 8 weeks, with all meals provided; (ii) controlled 7-10% weight loss with caloric intake reduced by 25% to achieve the desired amount of weight loss in about 4 to 5 months with all meals provided; and (iii) Independent weight loss for about 4 months. During the independent weight loss phase of the study subjects will be asked to continue to consume a plant-based, very-low-fat diet but will prepare all their food at home. No food will be provided during this portion of the study.
  Arms: Metabolically abnormal obese - Plant-based very-low-fat diet
Behavioral: Annual Follow-up Visits — Metabolic health will be assessed 1 and 2-years after competing the diet intervention study. No intervention will be performed during the time.
  Arms: Metabolically abnormal obese - Low carbohydrate ketogenic diet; Metabolically abnormal obese - Mediterranean diet; Metabolically abnormal obese - Plant-based very-low-fat diet

SUMMARY:
The purpose of this research study is to 1) understand how some, but not all people with obesity develop obesity related conditions such as type 2 diabetes and cardiovascular disease, and 2) compare the effects of 3 popular weight loss diets (Mediterranean, low-carbohydrate, or a very-low-fat plant-based diet) in people with obesity.

DETAILED DESCRIPTION:
Obesity is associated with a constellation of cardiometabolic abnormalities (including insulin resistance, elevated blood pressure and dyslipidemia) that are risk factors for diabetes and cardiovascular disease. However, not all people experience the typical "complications" associated with obesity. Approximately 25% of obese people are protected from the adverse metabolic effects of excess fat accumulation and are considered metabolically-normal, based on their normal response to insulin. The mechanisms responsible for the development of insulin resistance and cardiometabolic complications in some, but not all, obese persons are unknown.

In people that do develop the typical "complications" associated with obesity weight loss has profound therapeutic effects. Currently, there are three distinctly different types of diets that have demonstrated considerable benefits in improving cardiometabolic health in both lean and obese people: 1) a Mediterranean diet, 2) a low-carbohydrate, ketogenic diet, and 3) a plant-based, very-low-fat diet. However, there is considerable inter-individual variability in body weight loss among people in response to any given diet, and it is not known why some people lose more weight with one diet than another. The mechanisms responsible for the different weight and metabolic responses to specific types of diets and the independent effects of weight loss and dietary macronutrient composition on cardiometabolic health are unclear.

The overarching goal of this project is therefore to fill these gaps in knowledge by conducting a careful cross-sectional characterization of metabolically normal lean, metabolically normal obese and metabolically abnormal obese individuals to compare body composition, body fat distribution, the plasma metabolome, systemic and adipose tissue inflammation and immune system function, adipose tissue and muscle biological function, the gut microbiome, the brain's structure, cognitive function and central reward mechanisms, and taste sensation between groups. . Metabolically abnormal obese participants will then be randomized to follow a Mediterranean, a low-carbohydrate ketogenic or a plant-based, very-low-fat diet to examine the different effects of these diets on the above outcomes with the purpose to determine the beneficial or potentially harmful effects of these different diets.

ELIGIBILITY:
Inclusion Criteria:

* Metabolically normal lean subjects must have a BMI ≥18.5 and ≤24.9 kg/m2; Obese subjects must have a BMI ≥30.0 and ≤50.0 kg/m2
* Metabolically normal lean and obese subjects must have intrahepatic triglyceride (IHTG) content ≤5%; plasma triglyceride (TG) concentration <150 mg/dl; fasting plasma glucose concentration <100 mg/dl, 2-hr oral glucose tolerance plasma glucose concentration <140 mg/dl, and hemoglobin A1C ≤5.6%
* Metabolically abnormal obese subjects must have intrahepatic triglyceride (IHTG) content ≥5.6%; HbA1C ≥5.7%, or fasting plasma glucose concentration ≥100 mg/dl, or 2-hr oral glucose tolerance test (OGTT) plasma glucose concentration ≥140 mg/dl.

Exclusion Criteria:

* Medical, surgical, or biological menopause
* Previous bariatric surgery where the gastrointestinal tract is reconstructed such as Roux-en-Y, sleeve gastrectomy and biliopancreatic diversion surgeries
* Laparoscopic adjustable gastric band (lab band) surgery within the last 3 years
* Structured exercise ≥250 min per week (e.g., brisk walking)
* Unstable weight (>4% change during the last 2 months before entering the study)
* Significant organ system dysfunction (e.g., diabetes requiring medications, severe pulmonary, kidney or cardiovascular disease)
* Polycystic ovary syndrome
* Cancer or cancer that has been in remission for <5 years
* Major psychiatric illness
* Conditions that render subject unable to complete all testing procedures (e.g., severe ambulatory impairments, limb amputations, or metal implants that interfere with imaging procedures; coagulation disorders)
* Use of medications that are known to affect the study outcome measures (e.g., steroids, non-statin lipid-lowering medications) or increase the risk of study procedures (e.g., anticoagulants) and that cannot be temporarily discontinued for this study
* Use of antibiotics in last 60 days
* Smoke cigarettes > 10 cigarettes/week
* Use marijuana >2 x/week, or use of illegal drugs
* Men who consume >21 units (e.g. glass of wine or bottle of beer) of alcohol per week and women who consume >14 units of alcohol per week
* Pregnant or lactating women
* Vegans, vegetarians, those with lactose intolerance and/or severe aversions/sensitivities to eggs, fish, nuts, wheat and soy, and/or any individuals with food allergies that induce an anaphylactic response
* Persons who are not able to grant voluntary informed consent
* Persons who are unable or unwilling to follow the study protocol or who, for any reason, the research team considers not an appropriate candidate for this study, including non-compliance with screening appointments or study visits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-02; Primary Completion 2025-04 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Whole-body insulin sensitivity will be assessed by using the hyperinsulinemic-euglycemic clamp procedure
Change in insulin sensitivity | Before and after 4 to 8-weeks of weight maintenance and after 7-10% weight loss (~6-7 months)
  Whole-body insulin sensitivity will be assessed by using the hyperinsulinemic-euglycemic clamp procedure

SECONDARY OUTCOMES:
24-hour glucose concentrations | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Glucose concentrations will be evaluated from frequent blood samples over a 24 h period
Change in 24-hour glucose concentrations | Before and after 4 to 8-weeks of weight maintenance and after 7-10% weight loss (~6-7 months)
  Glucose concentrations will be evaluated from frequent blood samples over a 24 h period
24-hour hormone concentrations | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Plasma hormone concentrations will be evaluated from frequent blood sampling over a 24 h period
Change in 24-hour hormone concentrations | Before and after 4 to 8-weeks of weight maintenance and after 7-10% weight loss (~6-7 months)
  Plasma hormone concentrations will be evaluated from frequent blood sampling over a 24 h period
24-hour cytokine concentrations | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Plasma cytokine concentrations will be evaluated from frequent blood sampling over a 24 h period
β-cell function | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  β-cell function will be assessed from a modified oral glucose tolerance test
Change in β-cell function | Before and after 7-10% weight loss (~6-7 months) and independent weight loss (12 months) in metabolically abnormal obese individuals only.
  β-cell function will be assessed from a modified oral glucose tolerance test
Insulin clearance | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Insulin clearance will be assessed from a modified oral glucose tolerance test and hyperinsulinemic-euglycemic clamp procedure
Insulin clearance | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only.
  Insulin clearance will be assessed from a modified oral glucose tolerance test and hyperinsulinemic-euglycemic clamp procedure
Fat mass and fat free mass | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Change in fat mass and fat free mass | Before and after 4 to 8-weeks of weight maintenance, after 7-10% weight loss (~6-7 months) and after independent weight loss (12 months)
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Exosome-mediated intercellular signaling | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Signaling between cells and organs will be examined by isolating exosomes (small extracellular vesicles) from blood and adipose tissue
Change in exosome-mediated intercellular signaling | Before and after 4 to 8-weeks of weight maintenance, after 7-10% weight loss (~6-7 months) and after independent weight loss (12 months)
  Signaling between cells and organs will be examined by isolating exosomes (small extracellular vesicles) from blood and adipose tissue
Abdominal adipose tissue volumes | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Abdominal subcutaneous and intra-abdominal adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Change in abdominal adipose tissue volumes | Before and after 4 to 8-weeks of weight maintenance, after 7-10% weight loss (~6-7 months) and after independent weight loss (12 months)
  Abdominal subcutaneous and intra-abdominal adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Leg adipose tissue volumes | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Thigh and calf adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Change in leg adipose tissue volumes | Before and after 4 to 8-weeks of weight maintenance, after 7-10% weight loss (~6-7 months) and after independent weight loss (12 months)
  Thigh and calf adipose tissue volumes will be assessed by magnetic resonance imagining (MRI)
Intra-hepatic triglyceride content | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Intra-hepatic triglyceride content will be assessed by magnetic resonance techniques
Change in intra-hepatic triglyceride content | Before and after 4 to 8-weeks of weight maintenance, after 7-10% weight loss (~6-7 months) and after independent weight loss (12 months)
  Intra-hepatic triglyceride content will be assessed by magnetic resonance techniques
Gut microbiome | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Gut microbiota, meta-transcriptome (bacterial RNA sequencing to determine what proteins can be made by the microbiota) and the meta-metabolome (metabolites made by the microbiota) will be assessed
Change in gut microbiome | Before and during 4 to 8-weeks of weight maintenance, 7-10% weight loss (~6-7 months) and independent weight loss (12 months)
  Gut microbiota, meta-transcriptome (bacterial RNA sequencing to determine what proteins can be made by the microbiota) and the meta-metabolome (metabolites made by the microbiota) will be assessed
Plasma lipid profile | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Fasting plasma lipid profile will be assessed by nuclear magnetic resonance (NMR) techniques
Change in plasma lipid profile | Before and after 4 to 8-weeks of weight maintenance, after 7-10% weight loss (~6-7 months) and after independent weight loss (12 months)
  Fasting plasma lipid profile will be assessed by nuclear magnetic resonance (NMR) techniques
Aerobic fitness | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Maximal oxygen consumption will be assessed using indirect calorimetry during a graded exercise test to volitional fatigue
Change in aerobic fitness | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals randomized to the plant-based very-low-fat diet only
  Maximal oxygen consumption will be assessed using indirect calorimetry during a graded exercise test to volitional fatigue
Carotid artery intima media thickness | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Carotid artery intima media thickness will be assessed by ultrasound imaging
Change in carotid artery intima media thickness | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Carotid artery intima media thickness will be assessed by ultrasound imaging
Cardiac structure and function | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Ultrasound techniques will be used to assess cardiac structure and function
Change in cardiac structure and function | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Ultrasound techniques will be used to assess cardiac structure and function
Endothelial function | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Endothelial function will be assessed using a non-invasive device (EndoPat 2000) in response to reactive hyperemia.
Change in endothelial function | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Endothelial function will be assessed using a non-invasive device (EndoPat 2000) in response to reactive hyperemia.
Arterial stiffness | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Arterial stiffness will be assessed using a non-invasive device (SphygmoCor)
Change in arterial stiffness | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Arterial stiffness will be assessed using a non-invasive device (SphygmoCor)
Physical activity | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Physical activity will be assessed using tri-axial accelerometry
Change in physical activity | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Physical activity will be assessed using tri-axial accelerometry
Sleep efficiency | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Sleep efficiency will be assessed using tri-axial accelerometry
Change in sleep efficiency | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Sleep efficiency will be assessed using tri-axial accelerometry
Rate of incorporation of 2H2O into lipids | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Metabolic pathways relating to lipid (fat) synthesis in the liver and adipose tissue (fat) will be assessed by heavy water (2H2O) ingestion followed by fat biopsies and blood sampling
Change in the rate of incorporation of 2H2O into lipids | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Metabolic pathways relating to lipid (fat) synthesis in the liver and adipose tissue (fat) will be assessed by heavy water (2H2O) ingestion followed by fat biopsies and blood sampling
Rate of incorporation of 2H2O into proteins | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Metabolic pathways relating to protein synthesis in the muscle and adipose tissue will be assessed by heavy water (2H2O) ingestion followed by skeletal muscle and and adipose tissue biopsies and blood sampling
Change in the rate of incorporation of 2H2O into proteins | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Metabolic pathways relating to protein synthesis in the muscle and adipose tissue will be assessed by heavy water (2H2O) ingestion followed by skeletal muscle and and adipose tissue biopsies and blood sampling
Taste intensity | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Subjects will be evaluated by using the NIH toolbox Taste Intensity Test
Change in taste intensity | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Subjects will be evaluated by using the NIH toolbox Taste Intensity Test
Sweet taste palatability | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Sweet palatability will be assessed using the general Labeled Magnitude Scale
Change in sweet taste palatability | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Sweet palatability will be assessed using the general Labeled Magnitude Scale
Immune function | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Immune cell populations within plasma and adipose tissue will be profiled using multi-color fluorescence activated cell sorting (FACS) techniques.
Change in immune function | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Immune cell populations within plasma and adipose tissue will be profiled using multi-color fluorescence activated cell sorting (FACS) techniques.
Food consumption-induced changes in brain blood flow | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Food consumption-induced changes in brain blood flow will be assessed by blood-oxygen dependent (BOLD) and arterial spin labeling using functional magnetic resonance imaging (fMRI) techniques
Change in food consumption-induced changes in brain blood flow | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  Food consumption-induced changes in brain blood flow will be assessed by blood-oxygen dependent (BOLD) and arterial spin labeling using functional magnetic resonance imaging (fMRI) techniques
Transcriptome in blood, muscle and adipose tissue | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  The transcriptome (all RNA that are responsible for making proteins from DNA templates) will be evaluated by using RNA sequencing techniques
Change in transcriptome in blood, muscle and adipose tissue | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  The transcriptome (all RNA that are responsible for making proteins from DNA templates) will be evaluated by using RNA sequencing techniques
Epigenome in blood, muscle and adipose tissue | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  The epigenome (chemical modifications of DNA that signal genes to be on or off) will be evaluated by using Illumina Infinium HumanMethylation450 BeadChip assays.
Change in epigenome in blood, muscle and adipose tissue | Before and after 7-10% weight loss (~6-7 months) in metabolically abnormal obese individuals only
  The epigenome (chemical modifications of DNA that signal genes to be on or off) will be evaluated by using Illumina Infinium HumanMethylation450 BeadChip assays.
Dopamine receptor binding potential | Baseline in fasted and fed states in metabolically abnormal obese participants only.
  Dopamine receptor binding potential will be assessed by Positron Emission Tomography (PET) using [11C]raclopride in the fasted and fed states
Subcutaneous abdominal adipose tissue oxygen tension | Baseline only (cross-sectional comparison of metabolically normal lean, metabolically normal obese and metabolically abnormal obese subjects).
  Oxygen tension will be assessed in subcutaneous abdominal adipose tissue in the abdomen using oxygen-sensitive fiber-optic probes (OxyLiteTM, Oxford Optronix, Ltd)
Change in β-cell function | Before and at annual follow-up visits (assessed up to 2 years) in metabolically abnormal obese individuals only.
  β-cell function will be assessed from a modified oral glucose tolerance test
Insulin clearance | Before and at annual follow-up visits (assessed up to 2 years) in metabolically abnormal obese individuals only.
  Insulin clearance will be assessed from a modified oral glucose tolerance test
Change in fat mass and fat free mass | Before and at annual follow-up visits (assessed up to 2 years) in metabolically abnormal obese individuals only.
  Fat mass and fat free mass will be assessed using dual-energy x-ray absorptiometry (DXA)
Change in intra-hepatic triglyceride content | Before and at annual follow-up visits (assessed up to 2 years) in metabolically abnormal obese individuals only.
  Intra-hepatic triglyceride content will be assessed by magnetic resonance techniques

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Petersen MC, Smith GI, Palacios HH, Farabi SS, Yoshino M, Yoshino J, Cho K, Davila-Roman VG, Shankaran M, Barve RA, Yu J, Stern JH, Patterson BW, Hellerstein MK, Shulman GI, Patti GJ, Klein S. Cardiometabolic characteristics of people with metabolically healthy and unhealthy obesity. Cell Metab. 2024 Apr 2;36(4):745-761.e5. doi: 10.1016/j.cmet.2024.03.002. PMID 38569471
- [Background] Mittendorfer B, van Vliet S, Smith GI, Petersen MC, Patterson BW, Klein S. Impaired plasma glucose clearance is a key determinant of fasting hyperglycemia in people with obesity. Obesity (Silver Spring). 2024 Mar;32(3):540-546. doi: 10.1002/oby.23963. Epub 2024 Jan 16. PMID 38228469
- [Result] Seo JB, Riopel M, Cabrales P, Huh JY, Bandyopadhyay GK, Andreyev AY, Murphy AN, Beeman SC, Smith GI, Klein S, Lee YS, Olefsky JM. Knockdown of Ant2 Reduces Adipocyte Hypoxia And Improves Insulin Resistance in Obesity. Nat Metab. 2019 Jan;1(1):86-97. doi: 10.1038/s42255-018-0003-x. Epub 2018 Nov 19. PMID 31528845
- [Result] Stern JH, Smith GI, Chen S, Unger RH, Klein S, Scherer PE. Obesity dysregulates fasting-induced changes in glucagon secretion. J Endocrinol. 2019 Nov;243(2):149-160. doi: 10.1530/JOE-19-0201. PMID 31454790
- [Result] Eisenstein SA, Black KJ, Samara A, Koller JM, Dunn JP, Hershey T, Klein S, Smith GI. Striatal Dopamine Responses to Feeding are Altered in People with Obesity. Obesity (Silver Spring). 2020 Apr;28(4):765-771. doi: 10.1002/oby.22753. Epub 2020 Feb 21. PMID 32086877
- [Result] Ding X, Iyer R, Novotny C, Metzger D, Zhou HH, Smith GI, Yoshino M, Yoshino J, Klein S, Swaminath G, Talukdar S, Zhou Y. Inhibition of Grb14, a negative modulator of insulin signaling, improves glucose homeostasis without causing cardiac dysfunction. Sci Rep. 2020 Feb 25;10(1):3417. doi: 10.1038/s41598-020-60290-1. PMID 32099031
- [Result] Smith GI, Polidori DC, Yoshino M, Kearney ML, Patterson BW, Mittendorfer B, Klein S. Influence of adiposity, insulin resistance, and intrahepatic triglyceride content on insulin kinetics. J Clin Invest. 2020 Jun 1;130(6):3305-3314. doi: 10.1172/JCI136756. PMID 32191646
- [Result] Smith GI, Shankaran M, Yoshino M, Schweitzer GG, Chondronikola M, Beals JW, Okunade AL, Patterson BW, Nyangau E, Field T, Sirlin CB, Talukdar S, Hellerstein MK, Klein S. Insulin resistance drives hepatic de novo lipogenesis in nonalcoholic fatty liver disease. J Clin Invest. 2020 Mar 2;130(3):1453-1460. doi: 10.1172/JCI134165. PMID 31805015
- [Result] Cifarelli V, Beeman SC, Smith GI, Yoshino J, Morozov D, Beals JW, Kayser BD, Watrous JD, Jain M, Patterson BW, Klein S. Decreased adipose tissue oxygenation associates with insulin resistance in individuals with obesity. J Clin Invest. 2020 Dec 1;130(12):6688-6699. doi: 10.1172/JCI141828. PMID 33164985
- [Result] Beals JW, Smith GI, Shankaran M, Fuchs A, Schweitzer GG, Yoshino J, Field T, Matthews M, Nyangau E, Morozov D, Mittendorfer B, Hellerstein MK, Klein S. Increased Adipose Tissue Fibrogenesis, Not Impaired Expandability, Is Associated With Nonalcoholic Fatty Liver Disease. Hepatology. 2021 Sep;74(3):1287-1299. doi: 10.1002/hep.31822. Epub 2021 Jun 22. PMID 33743554
- [Result] Fuchs A, Samovski D, Smith GI, Cifarelli V, Farabi SS, Yoshino J, Pietka T, Chang SW, Ghosh S, Myckatyn TM, Klein S. Associations Among Adipose Tissue Immunology, Inflammation, Exosomes and Insulin Sensitivity in People With Obesity and Nonalcoholic Fatty Liver Disease. Gastroenterology. 2021 Sep;161(3):968-981.e12. doi: 10.1053/j.gastro.2021.05.008. Epub 2021 May 15. PMID 34004161
- [Result] Farabi SS, Smith GI, Schweitzer GG, Stein RI, Klein S. Do lifestyle factors and quality of life differ in people with metabolically healthy and unhealthy obesity? Int J Obes (Lond). 2022 Oct;46(10):1778-1785. doi: 10.1038/s41366-022-01180-6. Epub 2022 Jul 11. PMID 35817849
- [Result] Mittendorfer B, Patterson BW, Smith GI, Yoshino M, Klein S. beta Cell function and plasma insulin clearance in people with obesity and different glycemic status. J Clin Invest. 2022 Feb 1;132(3):e154068. doi: 10.1172/JCI154068. PMID 34905513
- [Result] Dunn JP, Lamichhane B, Smith GI, Garner A, Wallendorf M, Hershey T, Klein S. Dorsal striatal response to taste is modified by obesity and insulin resistance. Obesity (Silver Spring). 2023 Aug;31(8):2065-2075. doi: 10.1002/oby.23799. PMID 37475685
- [Result] Beals JW, Kayser BD, Smith GI, Schweitzer GG, Kirbach K, Kearney ML, Yoshino J, Rahman G, Knight R, Patterson BW, Klein S. Dietary weight loss-induced improvements in metabolic function are enhanced by exercise in people with obesity and prediabetes. Nat Metab. 2023 Jul;5(7):1221-1235. doi: 10.1038/s42255-023-00829-4. Epub 2023 Jun 26. PMID 37365374